CLINICAL TRIAL: NCT02805985
Title: Post-market Surveillance Study of FLXfit™ TLIF Interbody Fusion Device
Acronym: FLXFit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Expanding Orthopedics Ltd. (Industry)
Collaborators: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLXFit
Record Dates: First submitted 2016-05-25; First posted 2016-06-20 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Retrolisthesis
Keywords: Degenerative Disc Disease; Spondylolisthesis; Retrolisthesis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FLXfit™ TLIF Interbody Fusion Device (Experimental): The FLXfit™ is an expandable, articulated interbody fusion device (IBFD) used in conjunction with supplemental fixation to provide structural stability in skeletally mature individuals following total or partial discectomy.
  Interventions: Device: FLXfit™ TLIF Interbody Fusion Device

INTERVENTIONS:
Device: FLXfit™ TLIF Interbody Fusion Device — The FLXfit™ is an expandable, articulated interbody fusion device (IBFD) used in conjunction with supplemental fixation to provide structural stability in skeletally mature individuals following total or partial discectomy.

SUMMARY:
This study is a post-market clinical follow-up study. A post-market, prospective clinical trial will be conducted. The data collected from this study will serve the purpose of confirming safety and performance of the FLXfit™ implant.

DETAILED DESCRIPTION:
As detailed by Expanding Orthopedics Inc., the FLXfit™ is an expandable, articulated interbody fusion device (IBFD) used in conjunction with supplemental fixation to provide structural stability in skeletally mature individuals following total or partial discectomy.

The FLXfit™ is a unique titanium cage which articulates laterally as well as expands in height. This enables larger footprint support as well as restoration of disc height and lordotic angle correction. A bullet-nose design facilitates self-distraction and ease of insertion. The open architecture of the device allows it to be packed with autogenous bone graft.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-70 y/o)
* Male or Female
* With the following conditions of the lumbar spine as confirmed by advanced imaging (CT or MRI), who is a candidate for primary spinal fusion procedure according to acceptable criteria for such medical conditions:

  * Degenerative disc disease with up to Grade I spondylolisthesis
  * Spondylolisthesis
* Failure of at least 6-months conservative treatment
* BMI < 40
* Patient to approve no pregnancy during the 24 months of study and no participation in other studies in parallel to this one
* Ability to read, understand, and sign informed consent

Exclusion Criteria:

* Infection, local to the operative site
* Signs of local inflammation
* Fever or leukocytosis
* Pregnancy
* Significant mental disorder or condition that could compromise the patient's ability to remember and comply with preoperative and postoperative instructions (e.g. current treatment for a psychiatric/psychosocial disorder, senile dementia, Alzheimer's disease, traumatic head injury)
* Prior surgical procedure (with the exception of decompression only procedure) at the index level(s) using the desired operative approach
* Prior fusion procedure at an adjacent level
* Any other condition which would preclude the potential benefit of spinal implant surgery, such as the presence of tumors or congenital abnormalities, fracture local to the operating site, elevation of segmentation rate unexplained by other diseases, elevation of white blood count (WBC), or a marked left shift in the WBC differential count
* Neuromuscular disorder that would engender unacceptable risk of instability, implant fixation failure, or complications in postoperative care
* Active local infection in or near the operative region
* Active systemic infection and/or disease
* Severe osteoporosis or insufficient bone density, which in the medical opinion of the physician precludes surgery or contraindicates instrumentation
* Endocrine or metabolic disorders known to affect osteogenesis (e.g. Paget's disease, renal osteodystrophy, hypothyroidism)
* Systemic disease that requires the chronic administration of nonsteroidal anti-inflammatory or steroidal drugs
* Suspected or documented allergy or intolerance to implant's materials
* Symptomatic cardiac disease
* Patient unwilling to cooperate with postoperative instructions.
* Any case where the implant components selected for use would be too large or too small to achieve a successful result.
* Patient having inadequate tissue coverage over the operative site or inadequate bone stock or quality.
* Any patient in which implant utilization would interfere with anatomical structures or expected physiological performance.
* Prior fusion at the level to be treated.
* Back VAS < 4/10

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Safety/Adverse Events | Up to 24 months
  All adverse events will be assessed by incidence and time to resolution of postoperative device-related complications and serious adverse events/incidence and time to reoperation/incidence and time to revision. All perioperative adverse events will be noted. Information will be obtained from the operative note regarding blood loos, length of surgery, procedural details and complications. Postoperative events including nausea, vomiting, wound complications, thromboembolic events will be assessed.

SECONDARY OUTCOMES:
Disability | 24 months
  Obtaining improvement in Oswestry Disability Index (ODI) disease-specific questionnaire up to 24 months following the procedure, as compared to patient's baseline. Mean change in score of the ODI from baseline to 24 months postoperatively
Change in Disability | Up to 24 months
  Obtaining improvement in Oswestry Disability Index (ODI) disease-specific questionnaire up to 24 months following the procedure, as compared to patient's baseline. Mean change in score of the ODI from baseline to 24 months postoperatively
Pain | 24 months
  Obtaining improvement in Visual Analogue Scale (VAS) Back and Leg pain scores up to 24 months following the procedure as compared to patient's baseline. Mean change in score of the VAS from baseline to 24 months postoperatively
Change in Pain | Up to 24 months
  Obtaining improvement in Visual Analogue Scale (VAS) Back and Leg pain scores up to 24 months following the procedure as compared to patient's baseline. Mean change in score of the VAS from baseline to 24 months postoperatively
Health-Related Quality of Life Questionnaire | 24 months
  Obtaining improvement in Short Form-12 health survey up to 24 months following the procedure as compared to patient's baseline. Mean change in score of the SF-12 from baseline to 24 months postoperatively
Change in Health-Related Quality of Life Questionnaire | Up to 24 months
  Obtaining improvement in Short Form-12 health survey up to 24 months following the procedure as compared to patient's baseline. Mean change in score of the SF-12 from baseline to 24 months postoperatively
Arthrodesis (Fusion) | 6 months, 12 months, 24 months
  CT based fusion assessment at 6 months, 12 months, and 24 months
Radiographic Analysis (Global Lumbar Lordosis) | Immediate Postoperative, 6-week, 12-week, 6-month, 12-month, 24-month follow-up visits
  Immediate Postoperative, and at the 6-week, 12-week, 6-month, 12-month, 24-month follow-up visits assessing global lumbar lordosis (LL) at the level treated with the FLXfit device.
Radiographic Analysis (Segmental Lumbar Lordosis) | Immediate Postoperative, 6-week, 12-week, 6-month, 12-month, 24-month follow-up visits
  Immediate Postoperative, and at the 6-week, 12-week, 6-month, 12-month, 24-month follow-up visits assessing segmental lumbar lordosis (LL) at the level treated with the FLXfit device.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin H Massel, BS, Study Director — Rush University Medical Center; Benjamin C Mayo, BA, Study Director — Rush University Medical Center; Fady Hijji, BS, Study Director — Rush University Medical Center; Kern Singh, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center; Department of Orthopedic Surgery, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes